CLINICAL TRIAL: NCT01704014
Title: Intraoperative Floppy Iris Syndrome in Korean Patients Taking α1-Adrenergic Receptor Antagonists
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-01-034
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Intraoperative Floppy Iris Syndrome
Keywords: occurrence of

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- α1-ARA Group: All patients on α1-ARA(α1-adrenergic receptor antagonists) medication who underwent cataract surgeries.
- Control Group: Age and sex-matched control subjects

SUMMARY:
Intraoperative floppy iris syndrome (IFIS) is a recently described condition observed during cataract surgery. It has been hypothesized that irreversible atrophy of the iris dilator muscle associated with α1-adrenergic receptor antagonists (α1-ARA) is responsible for IFIS. However the prevalence of IFIS in Korean population is not reported. The purpose of this study is to evaluate the prevalence and clinical manifestations of IFIS in relation to iris anatomical change in Korean patients taking α1-ARA.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cataract
* korean patients

Exclusion Criteria:

* history of iridocyclitis, iris neovascularization, or prior iris surgery
* traumatic cataracts, zonular dialysis, or cataracts associated with ocular disease (e.g., uveitis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All korean patients who underwent cataract surgeries in Samsung Medical Center
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
occurrence of intraoperative floppy iris syndrome | intraoperative